CLINICAL TRIAL: NCT04057911
Title: A Trial of Non-invasive Stimulation in Cervical Dystonia
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Western University, Canada (Other)
Responsible Party: Principal Investigator, Mandar Jog, Professor, Western University, Canada
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 114198
Record Dates: First submitted 2019-08-09; First posted 2019-08-15 (Actual); Last update posted 2019-09-26 (Actual); Status verified 2019-09

CONDITIONS: Cervical Dystonia
Keywords: Cervical dystonia; Non-invasive stimulation
MeSH Terms: conditions — Torticollis

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Real NIBS (Experimental): In Real NIBS arm, active Noninvasive brain stimulation (NIBS) will be given for 20 mins.
  Interventions: Device: Active NIBS
- Sham NIBS (Sham Comparator): In Sham NIBS arm, sham Noninvasive brain stimulation (NIBS) will be given for 20 mins.
  Interventions: Device: Sham NIBS

INTERVENTIONS:
Device: Active NIBS — Cathodal noninvasive brain stimulation will be given for 20 mins.
  Arms: Real NIBS
Device: Sham NIBS — The electrode placement will be same, but the electric current will be ramped down 5 seconds after the beginning of the stimulation
  Arms: Sham NIBS

SUMMARY:
Cervical dystonia (CD) is a common movement disorder. Despite the optimization of botulinum toxin injection (BoNT-A) parameters including muscle selection and dosing, a significant proportion of patients report low levels of satisfaction, and a few of them develop resistance to therapy. The only options for such patients would be invasive therapy such as pallidotomy or pallidal deep brain stimulation. Currently, studies are going on the effectiveness of noninvasive neurostimulation in different neurological disorders. Transcranial Direct Current Stimulation (tDCS) or transcranial pulsed current stimulation (tPCS) are known to be safe non-invasive intervention with almost no side effects that can be used to provide complementary treatment. To detect the dysfunctional regions five min resting state quantitative EEG (qEEG) eyes closed will be recorded and analyzed each time before and after noninvasive stimulation. The investigators will evaluate the efficacy of acute noninvasive stimulation in those CD patients who are already on 3 monthly BoNT-A therapy but the effect of BoNT-A is wearing off in 8 weeks. Kinematics (static and dynamic movements) of neck movements will be recorded using established technology before and after stimulation.

DETAILED DESCRIPTION:
Cervical dystonia (CD) is the most common adult onset dystonia. Abnormal sensorimotor integration and maladaptive plasticity have been proposed as possible mechanisms. Currently, there is no definite way to assess and modify this dysfunctional network. Deep brain stimulation (DBS) is one possible way, but it is invasive and being used in highly selected patients. Intramuscular injections of botulinum toxin injection (BoNT-A) are successful. However, 30% patients discontinue due to lack of efficacy, side effects like muscle atrophy and dysphagia and the effect may wear off by week 8. Importantly, injections don't change the abnormal networks, as patients need life-long treatment.

Noninvasive brain stimulation (NIBS) is an evolving therapeutic option. Repetitive transcranial magnetic stimulation (rTMS) has already been used in network modulation in CD. Although effective, cost, lack of portability and side effects remain issues of rTMS. Portable, better tolerated and cheaper options using transcranial direct current stimulation (tDCS) in Parkinson's disease, dystonia, tremor, ataxia and transcranial pulsed current stimulation (tPCS) in Parkinson's disease are exciting new options. However, with these methods of NIS, many challenges remain - dysfunctional network localization, selecting parameters to use, providing adequate stimulation to alter the network consistently, maintain the therapeutic benefit chronically and have consistent adoption by the patient and clinician community. These variables make this exciting approach high risk, yet high yield if successful.

In this study, the investigators will use a new quantitative electroencephalography (qEEG) technique to first localize global network dysfunction in CD. Kinematic analysis of the biomechanics of CD will be recorded. The efficacy of acute NIBS will be evaluated in those CD patients who are already on 3 monthly BoNT-A therapy but the effect of BoNT-A is wearing off in 8 weeks.The effect will be measured using qEEG and kinematics pre and post stimulation.

Noninvasive stimulation will be delivered through a pair of saline-soaked (0.9% NaCl) surface sponge electrodes. Stimulation will be given for 20 mins, single session. For the sham condition, the electrode placement will be same, but the electric current will be ramped down in 5 seconds after the beginning of the stimulation.

Neurophysiological EEG signals will be recorded, eyes-closed, no-task, using g.Nautilus g.tec wireless system. The g.tech system uses earclip reference sensors. The subject will be in a quiet place with less light or electromagnetic perturbations. During the resting state recordings, patients are seated in a comfortable arm chair and will be instructed to keep relaxed, with their eyes closed for 5 mins.

A paired t test will be used to compare baseline data and post tPCS data. Descriptive analysis of the neurological examination findings will be provided.

ELIGIBILITY:
Inclusion Criteria:

* Patients with cervical dystonia who are already on 3 monthly BoNT-A therapy but the effect of BoNT-A is wearing off in 8 weeks.

Exclusion Criteria:

* Patients who have other issues like known structural etiology, that can aggravate cervical dystonia
* Patients who are not able to provide informed consent

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Estimated)
Dates: Start 2019-09 (Estimated); Primary Completion 2021-09 (Estimated); Study Completion 2021-10 (Estimated)

PRIMARY OUTCOMES:
Changes in Toronto Western Spasmodic Torticollis Rating Scale (TWSTRS). | 3 months
  Toronto Western Spasmodic Torticollis Rating Scale (TWSTRS) will be assessed before and after stimulation. This scale is used to assess the severity of cervical dystonia and the success of its treatment. A total score of 0 to 35 can be achieved; this is made up of various sub scores- maximal excursion, duration of neck deviation, effect of sensory tricks, shoulder elevation/anterior displacement, range of motion, time to maintain in neutral position.
Changes in Network fragmentation using Quantitative Electroencephalography (qEEG) | 3 months
  We will do network fragmentation by 5 mins of resting quantitative Electroencephalography (EEG), pre and post stimulation. All the frequency bands will be analyzed. The change of frequency bands leading to change in network fragmentation will plotted.
Kinematic changes in angular deviation and amplitude measures | 3 months
  Angular deviations will be calculated by degree of freedom angular bias from calibrated neutral position. Amplitude measures will be reported as root mean square values.

CONTACTS AND LOCATIONS:
Overall Officials: Mandar Jog, MD, Principal Investigator — London Health Sciences Centre
Locations (1):
- London Health Sciences Centre, London, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Bradnam LV, Frasca J, Kimberley TJ. Direct current stimulation of primary motor cortex and cerebellum and botulinum toxin a injections in a person with cervical dystonia. Brain Stimul. 2014 Nov-Dec;7(6):909-11. doi: 10.1016/j.brs.2014.09.008. Epub 2014 Oct 7. No abstract available. PMID 25440290
- [Background] Angelakis E, Liouta E, Andreadis N, Leonardos A, Ktonas P, Stavrinou LC, Miranda PC, Mekonnen A, Sakas DE. Transcranial alternating current stimulation reduces symptoms in intractable idiopathic cervical dystonia: a case study. Neurosci Lett. 2013 Jan 15;533:39-43. doi: 10.1016/j.neulet.2012.11.007. Epub 2012 Nov 10. PMID 23149130